CLINICAL TRIAL: NCT01424566
Title: A Two-part, Placebo-controlled, Study of the Safety and Efficacy of Sativex® Oromucosal Spray (Sativex®; Nabiximols) as Adjunctive Therapy in Relieving Uncontrolled Persistent Chronic Pain in Patients With Advanced Cancer, Who Have Inadequate Analgesia Even With Optimized Chronic Opioid Therapy.
Brief Title: A Two-Part Study of Sativex® Oromucosal Spray for Relieving Uncontrolled Persistent Pain in Patients With Advanced Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GWCA1103; 2010-022905-17 (EudraCT Number)
Record Dates: First submitted 2011-08-25; First posted 2011-08-29 (Estimated); Results first posted 2018-04-23 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Pain; Advanced Cancer
Keywords: Cancer pain; Opioid therapy; Inadequate analgesia; Optimized chronic opioid therapy
MeSH Terms: conditions — Pain; Cancer Pain | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nabiximols (Experimental): Nabiximols was self-administered by participants as a 100 microliter (μL) oromucosal spray in the morning and evening, up to a maximum of 10 sprays per day for 2 or 7 weeks. Nabiximols oromucosal spray contained delta-9-tetrahydrocannabinol (THC) (27 milligrams [mg]/milliliter [mL]):cannabidiol (CBD) (25 mg/mL), in ethanol:propylene glycol (50:50) excipients, with peppermint oil (0.05%)flavoring. Each 100 μL actuation delivered 2.7 mg THC and 2.5 mg CBD.
  Interventions: Drug: Nabiximols
- Placebo (GA-0034) (Placebo Comparator): Placebo was self-administered by participants as a 100 μL oromucosal spray in the morning and evening, up to a maximum of 10 sprays per day for 5 weeks. Placebo oromucosal spray contained ethanol:propylene glycol (50:50) excipients, with peppermint oil (0.05%) flavoring and colorings.
  Interventions: Drug: Placebo (GA-0034)

INTERVENTIONS:
Drug: Nabiximols
  Other Names: Sativex®
  Arms: Nabiximols
Drug: Placebo (GA-0034)
  Arms: Placebo (GA-0034)

SUMMARY:
The primary objective of this study was to evaluate the efficacy of nabiximols (Sativex®), compared with placebo, when used as an adjunctive measure in relieving uncontrolled persistent chronic pain (not breakthrough pain) in participants with advanced cancer, who had inadequate analgesia even with optimized chronic opioid therapy.

This multi-center study was conducted in two parts. All participants enrolled into the trial received nabiximols during one of two parts of the study, but they did not know which part.

Eligible participants were not required to stop any of their current treatments or medications.

DETAILED DESCRIPTION:
This 11-week, multi-center, placebo-controlled study aimed to determine the efficacy, safety and tolerability of nabiximols administered as an adjunctive treatment for 5 weeks, versus placebo, assessed by a 2-part, randomized withdrawal design. The first part of the study (Part A) was single-blind (participants) and the second part of the study (Part B) was randomized, double-blind. Eligible participants had advanced cancer, with a clinical diagnosis of cancer related pain which was not wholly alleviated by their current optimized opioid treatment.

Qualifying participants entered the study at screening and commenced a 5- to 14-day eligibility period. During this period, eligible participants had 3 consecutive days where pain severity remained within defined parameters, break-through opioid usage had not exceeded an average of 4 episodes per day, and maintenance opioid medication and dose had not changed. Eligible participants underwent nabiximols titration during a single-blind treatment period lasting 10 days, followed by 4 days of therapy at the titrated dose. Participants who demonstrated an improvement of 15% or more on the score of the pain numerical rating scale were advanced to Part B, where they were randomized 1:1 to nabiximols or placebo in a double-blind fashion. Participants then received study treatments at their self-titrated doses for 5 weeks. After the end of the 5-week treatment period, participants were offered the option of entering an open-label extension (OLE) study; participants who entered the OLE up to 7 days after study completion had their follow-up assessments performed on the same day as their first OLE study visit. Participants that did not enter the OLE study had a safety follow up visit 14 days after treatment completion, which could be via telephone.

ELIGIBILITY:
Inclusion Criteria (abbreviated):

* The participant had advanced cancer for which there is no known curative therapy
* The participant had a clinical diagnosis of cancer related pain, which was not alleviated with their current optimized opioid treatment
* The participant received an optimized maintenance dose of Step 3 opioid therapy, preferably with a sustained release preparation, but also allowing a regular maintenance dose of around the clock use of immediate release preparations
* The participant received a daily maintenance dose Step 3 opioid therapy of less than or equal to a total daily opioid dose of 500 mg/day of morphine equivalence (including maintenance and break-through opioids)
* The participant was using no more than one type of break-through opioid analgesia

Exclusion Criteria (abbreviated):

* Had any planned clinical interventions that would have affected their pain (for example, chemotherapy or radiation therapy where, in the clinical judgment of the investigator, these would be expected to affect pain)
* The participant was currently using or had used cannabis or cannabinoid-based medications within 30 days of study entry and was unwilling to abstain for the duration of the study
* Had experienced myocardial infarction or clinically significant cardiac dysfunction within the last 12 months or had a cardiac disorder that, in the opinion of the investigator would have put the participant at risk of a clinically significant arrhythmia or myocardial infarction
* Had significantly impaired renal function
* Had significantly impaired hepatic function
* Female participants of child-bearing potential and male participants whose partner was of child-bearing potential, unless willing to ensure that they or their partner used effective contraception, for example, oral contraception, double barrier, intra-uterine device, during the study and for three months thereafter (however, a male condom was not to be used in conjunction with a female condom as this may not have proven effective)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2012-06-29 (Actual); Primary Completion 2015-07-10 (Actual); Study Completion 2015-12-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (61):
- Australia (2):
  - East Melbourne
  - Parkville
- Bulgaria (3):
  - Shumen
  - Varna
  - Vratsa
- Germany (3):
  - Lünen
  - Stadtroda
  - Wetzlar
- Hungary (5):
  - Budapest
  - Deszk
  - Komárom
  - Nyíregyháza
  - Szikszó
- India (3):
  - Bangalore
  - Jaipur
  - Pune
- Israel (6):
  - Ashkelon
  - Beersheba
  - Haifa
  - Jerusalem
  - Ramat Gan
  - Ẕerifin
- Italy (3):
  - Garbagnate Milanese
  - Piacenza
  - Torino
- Lithuania (3):
  - Klaipėda
  - Šiauliai
  - Vilnius
- Poland (10):
  - Bydgoszcz
  - Czeladź
  - Gdansk
  - Gliwice
  - Kłodzko
  - Opole
  - Ostrowiec Świętokrzyski
  - Poznan
  - Warsaw
  - Włocławek
- Romania (9):
  - Alba Iulia
  - Baia Mare
  - Brăila
  - Bucharest
  - Focşani
  - Oradea
  - Satu Mare
  - Sibiu
  - Suceava
- Spain (5):
  - Cadiz
  - Granada
  - Madrid
  - Salamanca
  - Seville
- Taiwan (4):
  - Changhua
  - Taichung
  - Tainan
  - Taipei
- United Kingdom (5):
  - Bury St Edmunds
  - Edinburgh
  - Glasgow
  - Manchester
  - Norwich

REFERENCES:
- [Background] Fallon MT, Albert Lux E, McQuade R, Rossetti S, Sanchez R, Sun W, Wright S, Lichtman AH, Kornyeyeva E. Sativex oromucosal spray as adjunctive therapy in advanced cancer patients with chronic pain unalleviated by optimized opioid therapy: two double-blind, randomized, placebo-controlled phase 3 studies. Br J Pain. 2017 Aug;11(3):119-133. doi: 10.1177/2049463717710042. Epub 2017 May 17. PMID 28785408

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per the Statistical Analyses Plan, all randomized participants who received at least 1 dose of study drug were analyzed in the Intent to Treat (ITT) population as per randomized treatment group. Participants were included and analyzed according to the treatment group they were randomized to.
Groups:
- Single-blind Nabiximols: Nabiximols was self-administered by participants as a 100 microliter (μL) oromucosal spray in the morning and evening, up to a maximum of 10 sprays per day, for 2 weeks. Nabiximols oromucosal spray contained delta-9-tetrahydrocannabinol (THC) (27 milligrams [mg]/milliliter [mL]):cannabidiol (CBD) (25 mg/mL), in ethanol:propylene glycol (50:50) excipients, with peppermint oil flavoring. Each 100 μL actuation delivered 2.7 mg THC and 2.5 mg CBD.
- Double-blind Nabiximols: Nabiximols was self-administered by participants as a 100 μL oromucosal spray in the morning and evening, for 5 weeks, at the same level of dosing attained during the last 4 days of the single-blind period; however, the number of sprays could be decreased based upon tolerability throughout the study. Nabiximols oromucosal spray contained THC (27 mg/mL):CBD (25 mg/mL), in ethanol:propylene glycol (50:50) excipients, with peppermint oil flavoring. Each 100 μL actuation delivered 2.7 mg THC and 2.5 mg CBD. To enter the double-blind treatment period (Part B), participants had to achieve at least a 15% improvement in Numerical Rating Scale (NRS) pain scores during the single-blind treatment period (Part A).
- Double-blind Placebo (GA-0034): Placebo was self-administered by participants as a 100 μL oromucosal spray in the morning and evening for 5 weeks, at the same level of dosing attained during the last 4 days of the single-blind period; however, the number of sprays could be decreased based upon tolerability throughout the study. Placebo oromucosal spray contained ethanol:propylene glycol (50:50) excipients, with peppermint oil (0.05%) flavoring and colorings. To enter the double-blind treatment period (Part B), participants had to achieve at least a 15% improvement in NRS pain scores during the single-blind treatment period (Part A).
Period: Single-blind Treatment
Arm/Group | Single-blind Nabiximols | Double-blind Nabiximols | Double-blind Placebo (GA-0034)
Started | 406 | 0 (Participants were not enrolled in this arm in the single-blind period.) | 0 (Participants were not enrolled in this arm in the single-blind period.)
Received at Least 1 Dose of Study Drug | 404 (Two participants did not administer any study drug.) | 0 | 0
Single-blind Safety Population | 404 | 0 | 0
Met Randomization Criteria | 206 | 0 | 0
Completed | 206 | 0 | 0
Not Completed | 200 | 0 | 0
Not completed — Adverse Event | 71 | 0 | 0
Not completed — Withdrawal by Subject | 16 | 0 | 0
Not completed — Withdrawal by Investigator | 2 | 0 | 0
Not completed — Did Not Meet Inclusion Criteria | 108 | 0 | 0
Not completed — Met Exclusion Criteria | 1 | 0 | 0
Not completed — Did Not Administer Any Study Drug | 2 | 0 | 0
Period: Double-blind Treatment
Arm/Group | Single-blind Nabiximols | Double-blind Nabiximols | Double-blind Placebo (GA-0034)
Started | 0 (Participants were not enrolled in this arm in the double-blind period.) | 103 (Participants were not enrolled in this arm in the single-blind period.) | 103 (Participants were not enrolled in this arm in the single-blind period.)
Received at Least 1 Dose of Study Drug | 0 | 103 | 103
Randomized Safety Population | 0 | 103 | 103
ITT Population | 0 | 103 | 103
Completed | 0 | 78 | 88
Not Completed | 0 | 25 | 15
Not completed — Adverse Event | 0 | 21 | 13
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — Withdrawal by Investigator | 0 | 1 | 1
Not completed — Lack of Efficacy | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All participants who were randomized and received at least 1 dose of study drug. Two participants who were randomized in the single-blind treatment period did not administer any study drug.
Groups:
- Single-blind Nabiximols: Nabiximols was self-administered by participants as a 100 μL oromucosal spray in the morning and evening, up to a maximum of 10 sprays per day, for 2 weeks. Nabiximols oromucosal spray contained THC (27 mg/mL):CBD (25 mg/mL), in ethanol:propylene glycol (50:50) excipients, with peppermint oil flavoring. Each 100 μL actuation delivered 2.7 mg THC and 2.5 mg CBD.
Arm/Group | Single-blind Nabiximols
Number analyzed (Participants) | 406
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 177
  Male | 229

OUTCOME MEASURES:

1. Primary Outcome: Change From Randomization Baseline In Mean NRS Average Pain At End Of Treatment
Description: Participants indicated the level of pain experienced in the last 24 hours on an 11-point NRS, where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine." Change in mean NRS average pain was calculated as: End of Treatment NRS average pain score - Randomization (Part B) Baseline NRS average pain score. The participant's Randomization (Part B) baseline pain 0-10 NRS value was the mean over the last 4 consecutive days of the single-blind treatment period (Part A; pre-randomization). A negative value indicates an improvement in average pain score from Randomization (Part B) Baseline.
Time Frame: Randomization Baseline, End of Treatment (Day 36 of the double-blind period)
Population: The ITT Population included all participants who were randomized, received at least 1 dose of study drug, and had at least 1 efficacy endpoint. Participants were analyzed according to the treatment group they were randomized to.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Double-blind Nabiximols: Nabiximols was self-administered by participants as a 100 μL oromucosal spray in the morning and evening for 5 weeks, at the same level of dosing attained during the last 4 days of the single-blind period; however, the number of sprays could be decreased based upon tolerability throughout the study. Nabiximols oromucosal spray contained THC (27 mg/mL):CBD (25 mg/mL), in ethanol:propylene glycol (50:50) excipients, with peppermint oil flavoring. Each 100 μL actuation delivered 2.7 mg THC and 2.5 mg CBD. To enter the double-blind treatment period (Part B), participants had to achieve at least a 15% improvement in NRS pain scores during the single-blind treatment period (Part A).
Arm/Group | Double-blind Nabiximols | Double-blind Placebo (GA-0034)
Number analyzed (Participants) | 103 | 103
units on a scale | 0.5 (1.3) | 0.5 (1.6)
Statistical Analysis 1: Comparison: Double-blind Nabiximols vs Double-blind Placebo (GA-0034); Test type: Superiority; p = 0.9173, ANCOVA; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.42 to 0.38]

2. Secondary Outcome: Percent Improvement From Eligibility Baseline In Mean NRS Average Pain Score At End Of Treatment
Description: Participants indicated level of pain in the last 24 hours on an 11-point NRS, where a score of 0 was "no pain" and 10 was "pain as bad as you can imagine". Eligibility Baseline = mean score from the 3-day eligibility period. End of Treatment = mean score over last (up to) 4 days to the final pain score at End of Treatment or up until Day 36 of the double-blind period, whichever is earlier, or final score available (prematurely terminated).
  Percentage improvement from baseline (Imp%) was calculated as:
  Imp% = (Eligibility Baseline pain NRS mean - End of Treatment pain NRS mean)/Eligibility Baseline pain NRS mean * 100.
  For participants who died or withdrew due to disease progression, Imp% values were used. For participants who died or withdrew unrelated to disease progression before end of Week 5, Imp% was zero for participants whose Imp% value was positive and it was Imp% for participants whose Imp% value was not positive.
Time Frame: Eligibility Baseline, End of Treatment (Day 36 of the double-blind period)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percent improvement
Arm/Group | Double-blind Nabiximols | Double-blind Placebo (GA-0034)
Number analyzed (Participants) | 103 | 103
percent improvement | 33.3 [18.2 to 51.8] | 35.7 [18.8 to 51.3]

3. Secondary Outcome: Change From Randomization Baseline In Mean NRS Worst Pain At End Of Treatment
Description: Participants indicated the level of worst pain experienced in the last 24 hours on an 11-point NRS, where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine." Change in mean NRS worst pain was calculated as: End of Treatment NRS worst pain score - Randomization (Part B) Baseline NRS worst pain score. The participant's Randomization (Part B) baseline worst pain 0-10 NRS value was the mean over the last 4 consecutive days of the single-blind treatment period (Part A; pre-randomization). A negative value indicates an improvement in worst pain score from Randomization (Part B) Baseline.
Time Frame: Randomization Baseline, End of Treatment (Day 36 of the double-blind period)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-blind Nabiximols | Double-blind Placebo (GA-0034)
Number analyzed (Participants) | 103 | 103
units on a scale | 0.2 (1.4) | 0.5 (1.6)

4. Secondary Outcome: Change From Randomization Baseline In Mean Sleep Disruption NRS At End Of Treatment
Description: Participants indicated the level of sleep disruption experienced in the last 24 hours on an 11-point NRS, where a score of 0 indicated "did not disrupt sleep" and a score of 10 indicated "completely disrupted (unable to sleep at all)." Change in mean sleep disruption NRS was calculated as: End of Treatment sleep disruption NRS score - Randomization (Part B) Baseline sleep disruption NRS score. The participant's Randomization (Part B) baseline sleep disruption 0-10 NRS value was the mean over the last 4 consecutive days of the single-blind treatment period (Part A; pre-randomization). A negative value indicates an improvement in sleep disruption score from Randomization (Part B) Baseline.
Time Frame: Randomization Baseline, End of Treatment (Day 36 of the double-blind period)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-blind Nabiximols | Double-blind Placebo (GA-0034)
Number analyzed (Participants) | 103 | 103
units on a scale | 0.2 (1.3) | 0.5 (1.4)

5. Secondary Outcome: Subject Global Impression Of Change At Last Visit (Up To Day 36 Of The Double-blind Period)
Description: The Subject Global Impression of Change (SGIC) was used to assess the overall status of the participant related to their cancer pain, with the markers "very much improved, much improved, slightly improved, no change, slightly worse, much worse, or very much worse". The SGIC was assessed at Day 36 of the double-blind period or the day at which a participant's last evaluation was performed, such as in the case of early termination. Last visit refers to the last visit that a participant completed the assessment; this could be either Day 22 or Day 36 of the double-blind period.
Time Frame: Last Visit (up to Day 36 of the double-blind period)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Nabiximols | Double-blind Placebo (GA-0034)
Number analyzed (Participants) | 88 | 97
Participants
  Very Much Improved | 6 | 6
  Much Improved | 28 | 35
  Slightly Improved | 35 | 26
  No Change | 8 | 15
  Slightly Worse | 8 | 8
  Much Worse | 3 | 6
  Very Much Worse | 0 | 1

6. Secondary Outcome: Physician Global Impression Of Change At Last Visit (Up To Day 36 Of The Double-blind Period)
Description: The Physician Global Impression of Change (PGIC) was used by the treating physician (investigator/sub-investigator) to assess if there was any change in the general functional abilities of the participant since prior to commencement of study medication, with the markers: "very much worse, much worse, slightly worse, no change, slightly improved, much improved, very much improved". Last visit refers to the last visit that a participant completed the assessment; this could be either Day 22 or Day 36 of the double-blind period.
Time Frame: Last Visit (up to Day 36 of the double-blind period)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Nabiximols | Double-blind Placebo (GA-0034)
Number analyzed (Participants) | 90 | 97
Participants
  Very Much Improved | 7 | 7
  Much Improved | 22 | 30
  Slightly Improved | 37 | 25
  No Change | 11 | 20
  Slightly Worse | 4 | 12
  Much Worse | 8 | 3
  Very Much Worse | 1 | 0

7. Secondary Outcome: Patient Satisfaction Questionnaire At Last Visit (Up To Day 36 Of The Double-blind Period)
Description: The Patient Satisfaction Questionnaire (PSQ) was used to assess level of satisfaction of the participant with the study drug, with the markers "extremely satisfied, very satisfied, slightly satisfied, neutral, slightly dissatisfied, very dissatisfied, extremely dissatisfied". Last visit refers to the last visit that a participant completed the assessment; this could be either Day 22 or Day 36 of the double-blind period.
Time Frame: Last Visit (up to Day 36 of the double-blind period)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Nabiximols | Double-blind Placebo (GA-0034)
Number analyzed (Participants) | 89 | 97
Participants
  Extremely Satisfied | 5 | 5
  Very Satisfied | 30 | 38
  Slightly Satisfied | 35 | 28
  Neutral | 14 | 10
  Slightly Dissatisfied | 2 | 11
  Very Dissatisfied | 0 | 4
  Extremely Dissatisfied | 3 | 1

8. Secondary Outcome: Change From Randomization Baseline In Daily Total Opioid Use (Morphine Equivalent) At End Of Treatment
Description: The total daily opioid use (in morphine equivalence) was the sum of morphine equivalence of daily maintenance dose and break-through dose.
  Change in daily total opioid use was calculated as: End of Treatment daily total opioid use - Randomization (Part B) Baseline daily total opioid use. The participant's Randomization (Part B) baseline daily total opioid use value was the mean over the last 4 consecutive days of the single-blind treatment period (Part A; pre-randomization). A negative value indicates a decrease in use from Randomization (Part B) Baseline.
Time Frame: Randomization Baseline, End of Treatment (Day 36 of the double-blind period)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg (morphine equivalent)
Arm/Group | Double-blind Nabiximols | Double-blind Placebo (GA-0034)
Number analyzed (Participants) | 103 | 103
mg (morphine equivalent) | 9.0 (45.6) | 15.5 (75.9)

9. Secondary Outcome: Change From Randomization Baseline In Daily Maintenance Opioid Dose (Morphine Equivalent) At End Of Treatment
Description: The prescribed daily quantity of opioid maintenance dose was calculated as the product of dose per use and daily frequency of use. Participants were asked: "Have you used your maintenance dose painkiller today as prescribed?" If the participant answered "No" to the question, the daily opioid maintenance dose usage on that day was set to 0.
  Change in daily maintenance opioid dose was calculated as: End of Treatment daily maintenance opioid dose - Randomization (Part B) Baseline daily maintenance opioid dose. The participant's Randomization (Part B) baseline daily maintenance opioid dose value was the mean over the last 4 consecutive days of the single-blind treatment period (Part A; pre-randomization). A negative value indicates a decrease in dose from Randomization (Part B) Baseline.
Time Frame: Randomization Baseline, End of Treatment (Day 36 of the double-blind period)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg (morphine equivalent)
Arm/Group | Double-blind Nabiximols | Double-blind Placebo (GA-0034)
Number analyzed (Participants) | 103 | 103
mg (morphine equivalent) | 0.0 (11.0) | 8.5 (54.6)

10. Secondary Outcome: Change From Randomization Baseline In Daily Break-through Opioid Dose (Morphine Equivalent) At End Of Treatment
Description: Daily break-through opioid dose usage was calculated as the product of prescribed dose per use, and the number of uses per day. If participants took more than 1 different break-through opioid for more than 1 day, the sum of morphine equivalence dose usages for each break-through opioid was calculated for the summary.
  Change in daily break-through opioid dose was calculated as: End of Treatment daily break-through opioid dose - Randomization (Part B) Baseline daily maintenance opioid dose. The participant's Randomization (Part B) baseline daily break-through opioid dose value was the mean over the last 4 consecutive days of the single-blind treatment period (Part A; pre-randomization). A negative value indicates a decrease in dose from Randomization (Part B) Baseline.
Time Frame: Randomization Baseline, End of Treatment (Day 36 of the double-blind period)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg (morphine equivalent)
Arm/Group | Double-blind Nabiximols | Double-blind Placebo (GA-0034)
Number analyzed (Participants) | 103 | 103
mg (morphine equivalent) | 9.0 (50.7) | 7.0 (36.1)

11. Secondary Outcome: Change From Randomization Baseline In NRS Constipation At Last Visit (Up To Day 36 Of The Double-blind Period)
Description: Participants indicated level of constipation on an 11-point NRS, where a score of 0 was "no constipation", and 10 was "constipation as bad as you can imagine." Last visit refers to the last visit that a participant completed the assessment.
  Change in NRS constipation score was calculated as: Last Visit NRS constipation score - Randomization (Part B) Baseline NRS constipation score. The participant's Randomization (Part B) baseline constipation NRS value was the last evaluation (including unscheduled visits) in the single-blind treatment period (Part A) prior to the first dose of study drug in the double-blind treatment period (Part B). A negative value indicates improvement in condition from Randomization (Part B) Baseline.
Time Frame: Randomization Baseline, Last Visit (up to Day 36 of the double-blind period)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-blind Nabiximols | Double-blind Placebo (GA-0034)
Number analyzed (Participants) | 89 | 96
units on a scale | 0.0 (1.8) | -0.2 (2.2)

ADVERSE EVENTS:
Time Frame: Up to Day 43 of the double-blind period post-randomization
Groups:
- Single-blind Nabiximols: Nabiximols was self-administered by participants as a 100 μL oromucosal spray in the morning and evening, up to a maximum of 10 sprays per day, for 2 weeks. Nabiximols oromucosal spray contained THC (27 mg/mL):CBD (25 mg/mL), in ethanol:propylene glycol (50:50) excipients, with peppermint oil flavoring. Each 100 μL actuation delivered 2.7 mg THC and 2.5 mg CBD. Two participants did not receive study drug and are not included in the safety set.
Arm/Group | Single-blind Nabiximols | Double-blind Nabiximols | Double-blind Placebo (GA-0034)
Serious Adverse Events (participants affected / at risk) | 80/404 | 33/103 | 16/103
Other Adverse Events (participants affected / at risk) | 97/404 | 21/103 | 17/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single-blind Nabiximols (N=404) | Double-blind Nabiximols (N=103) | Double-blind Placebo (GA-0034) (N=103)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal Perforation (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Breakthrough Pain (General disorders) | 1 | 0 | 0
General Physical Health Deterioration (General disorders) | 2 | 0 | 0
Pain (General disorders) | 2 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Acute Hepatic Failure (Hepatobiliary disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 2 | 0 | 0
Meningitis Listeria (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0
Pneumonia Bacterial (Infections and infestations) | 1 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 3 | 0 | 0
ECG Signs of Myocardial Ischaemia (Investigations) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 0
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 41 | 28 | 11
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0
Hypoglycaemic Coma (Nervous system disorders) | 1 | 0 | 0
Nerve Root Compression (Nervous system disorders) | 1 | 0 | 0
Sedation (Nervous system disorders) | 1 | 0 | 0
Spinal Cord Compression (Nervous system disorders) | 2 | 0 | 0
Renal Failure Acute (Renal and urinary disorders) | 2 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Anaemia of Malignant Disease (Blood and lymphatic system disorders) | 0 | 0 | 1
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1
Catheter Site Cellulitis (Infections and infestations) | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0
Abdominal Sepsis (Infections and infestations) | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0
Peripheral Embolism (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single-blind Nabiximols (N=404) | Double-blind Nabiximols (N=103) | Double-blind Placebo (GA-0034) (N=103)
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 6 | 3
Nausea (Gastrointestinal disorders) | 25 | 0 | 0
Vomiting (Gastrointestinal disorders) | 21 | 0 | 0
Dizziness (Nervous system disorders) | 27 | 0 | 0
Somnolence (Nervous system disorders) | 46 | 6 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 5 | 6
Asthenia (General disorders) | 0 | 6 | 6
Weight Decreased (Investigations) | 0 | 7 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days